CLINICAL TRIAL: NCT06164574
Title: Distinct Survivals and Optimal Combination of Immunotherapy Plus Immunophenotype in Uncommon and 20ins EGFR-mut Lung Adenocarcinoma: a Retrospective Multi-center Study
Brief Title: Immunotherapy in Uncommon and 20ins EGFR-mut Lung Cancers
Status: Completed | Type: Observational
Sponsor: Haiquan Chen (Other)
Responsible Party: Sponsor-Investigator, Haiquan Chen, Director in the Department of Thoracic Surgery, FUSCC, Fudan University
Organization: Fudan University (Other)
Other Study IDs: ImmEGFR
Record Dates: First submitted 2023-11-29; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Survival Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survival analysis — Immunotheray responses and long-term survival were evaluated in classical and other EGFR-mutant lung adenocarcinomas

SUMMARY:
Immunotherapy effectiveness and optimal combination strategy in lung cancers with EGFR uncommon and 20ins mutations was unclear. Based on 627 lung adenocarcinoma patients harboring EGFR mutations and receiving immunotherapy, we reported that patients with EGFR uncommon mutations had better response to immunotherapy, than EGFR 19del/L858R or 20in mutations. Immunotherapy monotherapy or plus chemotherapy was identified as better combination strategy for EGFR uncommon or 20ins mutations, respectively. Higher tumor mutation burden, more M1 macrophage, less Tregs and M2 macrophages infiltration, but not PD-L1 expression was found to be associated with EGFR uncommon mutations, compared to EGFR 19del/L858R or 20in mutations. These findings revealed diverse response and optimal combination strategy of lung adenocarcinoma patients harboring EGFR mutation subtypes, promoting rethinking about current immunotherapy application and prolonging survivals of them.

ELIGIBILITY:
Inclusion Criteria:

1. age≥18 years,
2. advanced or recurrent LUAD confirmed by pathology,
3. harboring EGFR mutations confirmed by super amplification refractory mutation system (super-ARMS) or next-generation sequencing (NGS),
4. receiving anti-PD-(L)1 antibody therapy at least once,
5. Radiologically evaluable according to Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: EGFR-mutant LUAD patients receiving anti-PD-(L)1 therapies
Sampling Method: Non-Probability Sample
Enrollment: 627 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Tumor response | From date of initial treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Partial response, disease progression, and stable disease were defined according to the RECIST v1.1

SECONDARY OUTCOMES:
Progression-free survivals | 5 years
  Progression-free survivals were defined as the time from the initial treatment to the date of disease progression or death

CONTACTS AND LOCATIONS:
Locations (1):
- Chaoqiang Deng, Shanghai, Please Select, China

IPD SHARING:
Plan to Share IPD: Undecided